CLINICAL TRIAL: NCT01319760
Title: MINI-AMI: Minimizing INfarct Size With IMPELLA® 2.5 System Following PCI for Acute Myocardial Infarction
Brief Title: MINI-AMI: Minimizing Infarct Size With Impella 2.5 Following PCI for Acute Myocardial Infarction
Acronym: MINI-AMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in business priority
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MINI-AMI G100286
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-04

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Sham Comparator): Patients in the control arm will be treated with standard of care for post-PCI STEMI patients in accordance with the the 2004 ACC/AHA Guidelines for the Management of Patients with ST-elevation Myocardial Infarction.
  Interventions: Other: Standard of care (Control)
- Impella 2.5 (Experimental): 24 hours of support with the Impella 2.5 post-PCI for acute myocardial infarction.
  Interventions: Device: Impella 2.5 support

INTERVENTIONS:
Device: Impella 2.5 support — Patients enrolled in the Impella arm will receive 24 hours of post-PCI hemodynamic support using the Impella 2.5
  Other Names: Impella LP 2.5
  Arms: Impella 2.5
Other: Standard of care (Control) — Standard care for STEMI patients post-PCI from ACC/AHA Guidelines
  Arms: Standard of care

SUMMARY:
A prospective, randomized, controlled multi-site feasibility trial to assess the potential role of the IMPELLA® 2.5 System in reducing infarct size in patients with ST-elevation myocardial infarction (STEMI)

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate whether the adjunctive use of the IMPELLA® 2.5 System for 24 hours following primary PCI for STEMI has the potential to limit the infarction of at-risk myocardium compared to primary PCI with routine post-PCI care (standard of care). This study is a feasibility study. Therefore, the principal objective is to identify trends in cardiac magnetic resonance imaging (MRI)-based efficacy outcomes between the randomized treatment arms (Impella arm compared standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed Informed Consent
* Acute anterior STEMI with ≥2 mm of ST-segment elevation in 2 or more contiguous anterior leads or ≥ 4 mm in total in the anterior leads, OR, Large Inferior STEMI with ≥2 mm of ST-segment elevation in 2 or more inferior leads AND EITHER ≥1 mm ST-segment elevation in V1 OR ≥1 mm of ST-segment depression in ≥2 contiguous anterior leads (V1-V3)
* Primary PCI performed within 5 hours of the onset of symptoms
* Patient undergoing emergent primary PCI of one culprit lesion in one major native epicardial coronary vessel
* Successful revascularization of the culprit native coronary artery with TIMI Flow Grade of 3 at the end of PCI

Exclusion Criteria:

* Cardiac arrest requiring CPR within 24 hours prior to enrollment
* Current cardiogenic shock
* Left Bundle Branch Block (new or old)
* Atrial fibrillation
* Known history of prior MI
* Prior coronary artery bypass graft surgery
* Known mural thrombus in the left ventricle or contraindication to left ventriculography
* Presence of a mechanical aortic valve
* Documented presence of moderate to severe aortic stenosis or moderate to severe aortic insufficiency.
* Known history of severe kidney dysfunction.
* Known contraindication to MRI (implanted metallic or magnetically activated device; claustrophobia, inability to hold breath for 15 seconds).
* History of recent (within 1 month) stroke or TIA
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
* Administration of fibrinolytic therapy within 24 hours
* Known hypersensitivity or contraindication to any of the following: Heparin, pork or pork products; Aspirin, All of the following: Clopidogrel, Ticlopidine, Prasugrel
* Contrast media Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device.
* Severe peripheral arterial obstructive disease that would preclude the IMPELLA® System placement
* Requirement to treat two or more culprit vessels during primary PCI, or plan for staged coronary revascularization (PCI or CABG) within the next 30 days.
* Inability to place Impella within 6 hours of the onset of symptoms, should patient be randomized to this arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Moses, MD, Principal Investigator — Columbia Presbyterian; Ajay Kirtane, MD, Principal Investigator — Columbia Presbyterian

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five roll-in subjects were enrolled in the MINI-AMI feasibility study between September 14, 2011 and April 24, 2012. A total of 82 patients have been screened but not enrolled by participating sites during the study period. Five (5) sites participated in the MINI-AMI study.
Pre-assignment Details: The study experienced a very low enrollment rate (lower than expected). The study was terminated before the roll-in phase was completed. No data for primary or secondary endpoints were collected in this study
Groups:
- Control (Standard of Care PCI Without Using Impella): Patients in the control arm will be treated with standard of care for postPCI STEMI patients in accordance with the 2004 ACC/AHA Guidelines for the Management of Patients with STelevation Myocardia Infarction
- Experimental (PCI Preceded With Impella 2.5): Patients in this arm will be treated in accordance with standard of care, and in addition will receive 24 hours of support with the Impella 2.5 postPCI for acute myocardial infarction.
  Impella 2.5 support: Patients enrolled in the Impella arm will receive 24 hours of postPCI hemodynamic support using the Impella 2.5.
Period: Overall Study
Arm/Group | Control (Standard of Care PCI Without Using Impella) | Experimental (PCI Preceded With Impella 2.5)
Started | 0 (The study experienced a very low enrollment rate. the sponsor decided to stop the study.) | 5
Completed | 0 (The study experienced a very low enrollment rate. the sponsor decided to stop the study.) | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only three (3) sites enrolled in the roll in phase. A total of five (5) patients were enrolled before the study was closed out. Investigators at each site were asked to enroll two initial roll-in patients that will be treated with the IMPELLA® 2.5 System.These roll in patients were not to be part of the primary analysis.
Groups:
- Control: Patients in the control arm will be treated with standard of care for post-PCI STEMI patients in accordance with the the 2004 ACC/AHA Guidelines for the Management of Patients with ST-elevation Myocardial Infarction.
  Control: Standard care for STEMI patients post-PCI from ACC/AHA Guidelines
- Impella 2.5: Patients in this arm will be treated in accordance with standard of care, and in addition will receive 24 hours of support with the Impella 2.5 post-PCI for acute myocardial infarction.
  Impella 2.5 support: Patients enrolled in the Impella arm will receive 24 hours of post-PCI hemodynamic support using the Impella 2.5
- Total: Total of all reporting groups
Arm/Group | Control | Impella 2.5 | Total
Number analyzed (Participants) | 0 | 5 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 61.8 (10.9) | 61.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 | 2
  Male |  | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Infarct Size
Description: Infarct size (as assessed by cardiac MRI at 3-5 days following the infarction).
Time Frame: 3-5 Days post infarct
Population: No data for primary or secondary endpoints were collected in this study
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Primary Outcome: No Data for Primary or Secondary Enpoints Were Collected
Time Frame: No data for primary or secondary enpoints were collected
Population: No data from primary or secondary endpoints were collected in this study
Groups:
- Roll In: Infarct size
Arm/Group | Roll In
Number analyzed (Participants) | 0

3. Secondary Outcome: Infarct Size
Description: Assessment of infarct size and remodeling characteristics at 90 days post-infarct.
Time Frame: 90 Days
Population: No data for primary or secondary endpoints were collected in this study
Groups:
- Roll in: Study close in roll in phase. therefore, no comparison data available.
Arm/Group | Roll in
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 90 days
Description: Study close in roll in phase. Therefore, no comparison data available.
Arm/Group | Roll In
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll In (N=5)
Decrease in Hemolobin (Blood and lymphatic system disorders) | 2 (2) — Bleeding
Cardiac Arrest (Cardiac disorders) | 1 (1) — Mortality (Cardiovascular and Non-cardiovascular)
Cardiogenic Shock (Vascular disorders) | 1 (1) — Vascular complications(sub-categorized as either Major or Minor)
chest pain (Cardiac disorders) | 1 (1)
Acute renal dysfunction (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll In (N=5)
Bleeding (Blood and lymphatic system disorders) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Significant platelet dysfunction (Blood and lymphatic system disorders) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2)
Worsening heart failure (Cardiac disorders) | 1 (1)
Acute Renal Dysfunction (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Study close in roll in phase. Therefore, no comparison data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No